CLINICAL TRIAL: NCT00441246
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter, Placebo-Controlled Study of the Safety and Efficacy of Mucinex D as Adjunct Therapy to Antibiotic Treatment of Acute Respiratory Infection
Brief Title: Phase 4 Study - Mucinex D as Adjunct Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adams Respiratory Therapeutics (Industry)
Responsible Party: Timothy Shea, Adams RT
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-MUCD-001
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Acute Respiratory Infection; Bronchitis; Rhinosinusitis
Keywords: Acute Respiratory Infection; Bronchitis; Rhinosinusitis
MeSH Terms: conditions — Bronchitis; Rhinosinusitis | interventions — Amiloride; Guaifenesin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Mucinex D (600 mg guaifenesin and 60 mg pseudoephedrine HCl extended-release bi-layer tablets)

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of Mucinex D tablets in providing symptom relief when administered as an adjunct to antibiotic therapy in patients with acute respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 to 75 years,
* Genders Eligible for Study: Both
* Adult patients presenting at the physician's office with symptoms diagnostic for acute respiratory infection, such as bronchitis or rhinosinusitis; with a clinical diagnosis of acute respiratory infection, meeting the physician's usual diagnostic criteria in practice for prescription of oral antibiotics.
* The investigator will evaluate patients on a total of seven criteria for inclusion.

Exclusion Criteria:

* Have chronic, recurring respiratory signs and symptoms, such as allergic rhinitis or chronic bronchitis, which, in the investigator's opinion, would confound interpretation of symptoms ratings for the acute respiratory infection;
* The Investigator will evaluate patients on twelve additional criteria for exclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The objective of the study is to evaluate the safety and efficacy of Mucinex D tablets in providing symptom relief when administered as an adjunct to antibiotic therapy in patients with acute respiratory infection. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Albrecht, M.D., Study Chair — Adams Respiratory Therapeutics
Locations (28):
- United States (28):
  - Alabama Clinical Therapuetics, LLC, 52 Medical Park East Drive, Suite 214, Birmingham, Alabama
  - MedCenter, 6651 Madison Ave., Carmichael, California
  - Torrance Clinical Research, 3640 Lomita Blfd #205, Torrance, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Longmont Clinic, P.C., 1925 W. Mountain View Ave., Longmont, Colorado
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - Dawsonville Family Medicine Clinical Trials, 5983 Hwy, 53E. Ste 175, Dawsonville, Georgia
  - Koch Family Medicine, 81A E. Queenwood Rd., Morton, Illinois
  - Welborn Clinic Gateway, 4233 Gateway Blvd, Newburgh, Indiana
  - Sterling Research Group, Ltd., 650 Sprucewood Lane, Erlanger, Kentucky
  - Columbia Medical Practice, 3450 Knoll Dr. North #200C, Columbia, Maryland
  - Clinical Associates, 750 Main St. #201, Reisterstown, Maryland
  - Milford Emergency Associates, Inc., 14 Asylum St., Milford, Massachusetts
  - Michigan Institute of Medicine, 38525 Eight Mile Rd., Livonia, Michigan
  - Central Nebraska Medical Clinic, PC, 145 Memorial Drive, Broken Bow, Nebraska
  - Immedicenter, 557 Broad St., Bloomfield, New Jersey
  - Central New York Clinical Research, RT 92, The Market Place, Manlius, New York
  - North Carolina Clinical Research, 4301 Lake Boone Trail, Ste 309-A, Raleigh, North Carolina
  - DayStar Clinical Research, Inc., 880 Mull Ave., Suite 100, Akron, Ohio
  - DataPharm, Inc., 6715 Tippecanoe Rd., Bldg E (LL), Canfield, Ohio
  - Parsons Avenue Medical Clinic, 1493 Parsons Avenue, Columbus, Ohio
  - Blair Medical Associates, Inc., Station Medical Center, 1414 Ninth Ave., Altoona, Pennsylvania
  - Harleysville Medical Associates, 176 Main Street, Harleysville, Pennsylvania
  - Lederach Family Medicine, PC, 658 Harleysville Pike, Suite 120, Harleysville, Pennsylvania
  - Greentree Medical Associates, 651 Holiday Drive, Foster Plaza Bldg #5, Pittsburgh, Pennsylvania
  - MetaClin Research, Inc., 6012 West William Cannon Drive, 6012 West William Cannon Drive, Austin, Texas
  - Apollo Research Institute, 117 Dilworth Plaza, Poth, Texas
  - Advanced Clinical Research, Inc., 3590 West 9000 South, Suite 230, West Jordan, Utah